CLINICAL TRIAL: NCT06973772
Title: Phase 3b, Multicenter, Randomized, Controlled, Double-Blind Clinical Trial to Evaluate the Immunogenicity and Safety of the Co-administration of Live Attenuated Dengue and Chikungunya Vaccines in Adults Aged 18 to 59 Years.
Brief Title: Trial to Evaluate the Immunogenicity and Safety of the Co-administration of Live Attenuated Dengue and Chikungunya Vaccines Compared to Separate Administration in Adults Aged 18 to 59 Years.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CODENCHIK-01-IB
Record Dates: First submitted 2025-04-28; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Dengue; Chikungunya
Keywords: dengue; chikungunya; coadministration regimen
MeSH Terms: conditions — Dengue; Chikungunya Fever | interventions — Vaccines, Attenuated; Vaccines

STUDY DESIGN:
Intervention Model Description: Phase 3b Multicenter, Randomized, Controlled, Double-Blind Clinical Trial to Evaluate the Immunogenicity and Safety of the Co-administration of Live Attenuated Dengue and Chikungunya Vaccines Compared to Separate Administration.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To ensure blinding of both participants and the study team performing safety assessments, vaccine preparation will be conducted by unblinded team members in a separate room, following the four-eyes principle (two individuals supervising the process). The syringes for different vaccination regimens will be pre-masked before being delivered to the study sites, ensuring the blinding process is maintained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dengue and Chikungunya vaccines co-administered (Experimental): A single dose of Butantan-DV + a single dose of VLA1555, administered concomitantly in opposite arms on Day 1.
  Interventions: Biological: DENGUE: Dengue 1,2,3,4 (attenuated) vaccine CHIKUNGUNYA: Chikungunya (CHIKV) live attenuated vaccine (VLA1555)
- Dengue vaccine only (Experimental): A single dose of Butantan-DV + placebo, administered concomitantly in opposite arms on Day 1.
  Interventions: Biological: DENGUE: Dengue 1,2,3,4 (attenuated) vaccine
- Chikungunya vaccine only (Experimental): A single dose of VLA1555 + placebo, administered concomitantly in opposite arms on Day 1.
  Interventions: Biological: Chikungunya (CHIKV) live attenuated vaccine (VLA1555)

INTERVENTIONS:
Biological: DENGUE: Dengue 1,2,3,4 (attenuated) vaccine CHIKUNGUNYA: Chikungunya (CHIKV) live attenuated vaccine (VLA1555) — DENGUE: Dose 10^2.5-4.1 PFU per virus (1,2,3,4) Route: Subcutaneous CHIKUNGUNYA: Dose >= 3.0 log TCID50 per 0.5 mL Route: Intramuscular
  Arms: Dengue and Chikungunya vaccines co-administered
Biological: DENGUE: Dengue 1,2,3,4 (attenuated) vaccine — DENGUE: Dose 10^2.5-4.1 PFU per virus (1,2,3,4) Route: Subcutaneous
  Arms: Dengue vaccine only
Biological: Chikungunya (CHIKV) live attenuated vaccine (VLA1555) — CHIKUNGUNYA: Dose >= 3.0 log TCID50 per 0.5 mL Route: Intramuscular
  Arms: Chikungunya vaccine only

SUMMARY:
This randomized, controlled, double blind trial aims at assessing the safety and immunogenicity profiles of the co-administered Live Attenuated Dengue and Chikungunya vaccines comparatively to the isolated administration, in the adult population aged 18 to 59 years without prior exposure to either arbovirus.

DETAILED DESCRIPTION:
A Phase 3b multicenter, randomized, controlled, double-blind clinical trial was designed to evaluate the Immunogenicity (non-inferiority), 28 days post-immunization, for each Dengue and Chikungunya serotypes, as well as the safety, 21 days post-immunization, of the co-administration of the live attenuated Dengue and Chikungunya vaccines compared to the separate administration in adults aged 18 to 59 years without prior exposure to either arbovirus.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18 to 59 years at the time of vaccination.
2. Signed informed consent by the participant or their legal representatives.
3. Ability to understand, based on the investigator's assessment, and agree to comply with all study procedures, including blood collection.

Exclusion Criteria:

1. Participation in another clinical trial within 28 days prior to screening or planned participation in another clinical study during the trial period.
2. Pre-existing unstable health condition. An unstable health condition is defined as a disease requiring a change in treatment or hospitalization due to disease worsening within 90 days prior to screening.
3. Vaccination within 14 days prior to screening with any inactivated vaccine or within 28 days prior to screening with any live attenuated vaccine, or planned vaccination with any vaccine up to 28 days after study vaccination.
4. Known hypersensitivity to any component of the vaccines.
5. Thrombocytopenia or bleeding disorders that contraindicate intramuscular vaccination or venipuncture for blood collection.
6. Receipt of immunoglobulins, blood, or blood products within 180 days prior to screening.
7. Altered immunocompetence (immunosuppression, immunodeficiency, or immunocompromise) primary or secondary due to: Clinical conditions (including but not limited to renal failure, liver failure with cirrhosis, heart failure class III or IV according to the New York Heart Association, HIV infection, and asplenia).
8. Use of systemic corticosteroids (oral, intravenous, or intramuscular) at a dose equivalent to ≥20 mg/day of prednisone for more than 14 days or a cumulative dose greater than 280 mg within the last 90 days prior to screening. Topical, inhaled, and intranasal corticosteroids are allowed. Intermittent use (a single dose within the last 30 days prior to screening) of intra-articular corticosteroids is also allowed.
9. Receipt of antineoplastic agents, immunosuppressants, immunomodulators, or radiotherapy within the last 180 days prior to screening.
10. Malignancy at the time of screening or a history of malignancy with <5 years of disease-free status at screening (except for basal cell carcinoma of the skin and localized prostate cancer under active surveillance).
11. Abuse of alcohol and illicit drugs within the past 12 months before screening that may compromise study compliance, at the investigator's discretion.
12. Being part of the study team, having a first-degree relative (parents, children, in-laws, stepchildren, sons-in-law, or daughters-in-law) or living in the same household as a study team member.
13. Any other clinical condition that, in the investigator's opinion, may interfere with the study results or pose an additional risk to the participant due to study inclusion.
14. Prior exposure to dengue and chikungunya viruses, i.e., non-reactive IgM and IgG as screened by specific ELISA for both viruses. In case of doubt or indeterminate ELISA results, at least two consecutive samples will be collected. If doubt persists after two test collections, the participant will be excluded.
15. For female participants of childbearing potential: Pregnancy (confirmed by a positive β-hCG test), breastfeeding, or intention to engage in sexual activity with reproductive potential without using a contraceptive method for 90 days following vaccination.
16. Previous receipt of any dengue or chikungunya vaccine.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity Primary | 28 days post-immunization
  Demonstrate the non-inferiority of the antibody response of co-administered Dengue and Chikungunya vaccines compared to Dengue and Chikungunya vaccines administered separately, for each Dengue serotype and Chikungunya in the adult population aged 18 to 59 years without prior exposure to either arbovirus, by calculating the Geometric Mean Titer (GMT) and the GMT ratio, post-immunization for each dengue serotype and chikungunya, across all intervention groups.
Safety Primary | 21 days post-immunization
  Assess the safety profile of co-administered Dengue and Chikungunya vaccines and Dengue and Chikungunya vaccines administered separately, in the adult population aged 18 to 59 years without prior exposure to either arbovirus, through the frequency of participants with solicited (local and systemic) and unsolicited adverse events (AEs), in all intervention groups.

SECONDARY OUTCOMES:
Immunogenicity Secondary 1 | 28 days post-immunization
  Assess the antibody response of co-administered Dengue and Chikungunya vaccines compared to Dengue and Chikungunya vaccines administered separately, in adults aged 18 to 59 years without prior exposure to either arbovirus, comparing the seroconversion rates, for each dengue serotype and chikungunya, across all intervention groups.
Immunogenicity Secondary 2. | 180 days post-immunization.
  Assess the antibody response of co-administered Dengue and Chikungunya vaccines compared to Dengue and Chikungunya vaccines administered separately, in adults aged 18 to 59 years without prior exposure to either arbovirus, comparing the Geometric Mean Titer and the GMT ratio, for each dengue serotype and chikungunya, across all intervention groups.
Safety Secondary 1. | up to 21 days post-immunization.
  Describe and compare the safety profile, by listing the Adverse Events of the co-administered Dengue and Chikungunya vaccines and Dengue and Chikungunya vaccines administered separately, reported in adults aged 18 to 59 years without prior exposure to either arbovirus.
Safety Secondary 2. | 180 days post-immunization
  Describe and compare the safety profile by listing Adverse Events of the co-administered Dengue and Chikungunya vaccines and Dengue and Chikungunya vaccines administered separately, in adults aged 18 to 59 years without prior exposure to either arbovirus.
Safety Secondary 3. | Days 1, 6, 9, 16, and 22.
  Describe post-vaccination viremia cases (manifestations).

CONTACTS AND LOCATIONS:
Locations (7):
- Brazil (7):
  - Centro Médico de São Francisco, Curitiba, Paraná
  - Centro de Pesquisa Inova, Toledo, Paraná
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Escola da Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul
  - Reumacenter, Porto Alegre, Rio Grande do Sul
  - UBEA - União Brasileira de Educação e Assistência Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa em AIDS do Estado do Rio Grande do Sul - IPARGS, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wressnigg N, Hochreiter R, Zoihsl O, Fritzer A, Bezay N, Klingler A, Lingnau K, Schneider M, Lundberg U, Meinke A, Larcher-Senn J, Corbic-Ramljak I, Eder-Lingelbach S, Dubischar K, Bender W. Single-shot live-attenuated chikungunya vaccine in healthy adults: a phase 1, randomised controlled trial. Lancet Infect Dis. 2020 Oct;20(10):1193-1203. doi: 10.1016/S1473-3099(20)30238-3. Epub 2020 Jun 1. PMID 32497524
- [Background] Schneider M, Narciso-Abraham M, Hadl S, McMahon R, Toepfer S, Fuchs U, Hochreiter R, Bitzer A, Kosulin K, Larcher-Senn J, Mader R, Dubischar K, Zoihsl O, Jaramillo JC, Eder-Lingelbach S, Buerger V, Wressnigg N. Safety and immunogenicity of a single-shot live-attenuated chikungunya vaccine: a double-blind, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 24;401(10394):2138-2147. doi: 10.1016/S0140-6736(23)00641-4. Epub 2023 Jun 12. PMID 37321235
- [Background] Nogueira ML, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, de Oliveira Alves LB, Infante V, Silveira DHR, de Lacerda MVG, Pereira DB, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Boaventura VS, Ramos F, Junior EE, de Moraes JC, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Kallas EG; Phase 3 Butantan-DV Working Group. Efficacy and safety of Butantan-DV in participants aged 2-59 years through an extended follow-up: results from a double-blind, randomised, placebo-controlled, phase 3, multicentre trial in Brazil. Lancet Infect Dis. 2024 Nov;24(11):1234-1244. doi: 10.1016/S1473-3099(24)00376-1. Epub 2024 Aug 5. PMID 39116904
- [Background] Kallas EG, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, Infante V, Palacios R, de Lacerda MVG, Batista Pereira D, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Barral AMP, Boaventura VS, Ramos F, Elias Junior E, Cassio de Moraes J, Covas DT, Kalil J, Precioso AR, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Nogueira ML. Live, Attenuated, Tetravalent Butantan-Dengue Vaccine in Children and Adults. N Engl J Med. 2024 Feb 1;390(5):397-408. doi: 10.1056/NEJMoa2301790. PMID 38294972
- [Background] Kallas EG, Precioso AR, Palacios R, Thome B, Braga PE, Vanni T, Campos LMA, Ferrari L, Mondini G, da Graca Salomao M, da Silva A, Espinola HM, do Prado Santos J, Santos CLS, Timenetsky MDCST, Miraglia JL, Gallina NMF, Weiskopf D, Sette A, Goulart R, Salles RT, Maestri A, Sallum AME, Farhat SCL, Sakita NK, Ferreira JCOA, Silveira CGT, Costa PR, Raw I, Whitehead SS, Durbin AP, Kalil J. Safety and immunogenicity of the tetravalent, live-attenuated dengue vaccine Butantan-DV in adults in Brazil: a two-step, double-blind, randomised placebo-controlled phase 2 trial. Lancet Infect Dis. 2020 Jul;20(7):839-850. doi: 10.1016/S1473-3099(20)30023-2. Epub 2020 Mar 24. PMID 32220283
- [Background] Chen LH, Fritzer A, Hochreiter R, Dubischar K, Meyer S. From bench to clinic: the development of VLA1553/IXCHIQ, a live-attenuated chikungunya vaccine. J Travel Med. 2024 Oct 19;31(7):taae123. doi: 10.1093/jtm/taae123. PMID 39255380
- [Background] Bonanni P, Steffen R, Schelling J, Balaisyte-Jazone L, Posiuniene I, Zatonski M, Van Damme P. Vaccine co-administration in adults: An effective way to improve vaccination coverage. Hum Vaccin Immunother. 2023 Dec 31;19(1):2195786. doi: 10.1080/21645515.2023.2195786. Epub 2023 Apr 11. PMID 37039318